CLINICAL TRIAL: NCT01099449
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind Study of Intravenous Calcium/Magnesium in Two Different Versions to Prevent Oxaliplatin-Induced Sensory Neurotoxicity
Brief Title: Calcium Gluconate and Magnesium Sulfate in Preventing Neurotoxicity in Patients With Colon Cancer or Rectal Cancer Receiving Oxaliplatin-Based Combination Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N08CB; NCCTG-N08CB; CDR0000669660 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02036 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Chemotherapeutic Agent Toxicity; Colorectal Cancer; Neuropathy; Neurotoxicity
Keywords: neurotoxicity; neuropathy; chemotherapeutic agent toxicity; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes; Colonic Neoplasms; Rectal Neoplasms | interventions — Calcium Gluconate; Magnesium Sulfate; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).
  Interventions: Drug: calcium gluconate; Drug: magnesium sulfate; Drug: oxaliplatin
- Arm II (Placebo Comparator): Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).
  Interventions: Other: placebo; Drug: oxaliplatin
- Arm III (Experimental): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).
  Interventions: Drug: calcium gluconate; Drug: magnesium sulfate; Other: placebo; Drug: oxaliplatin

INTERVENTIONS:
Drug: calcium gluconate — Given IV
  Arms: Arm I; Arm III
Drug: magnesium sulfate — Given IV
  Arms: Arm I; Arm III
Other: placebo — Given IV
  Arms: Arm II; Arm III
Drug: oxaliplatin

SUMMARY:
RATIONALE: Chemoprotective drugs, such as calcium gluconate and magnesium sulfate, may prevent neurotoxicity caused by oxaliplatin. It is not yet known which administration schedule of calcium gluconate and magnesium sulfate is more effective in preventing neurotoxicity.

PURPOSE: This randomized phase III trial is studying different administration schedules of calcium gluconate and magnesium sulfate and comparing how well they work in neurotoxicity in patients with colon cancer or rectal cancer receiving oxaliplatin-based combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether 2 schedules of calcium gluconate and magnesium sulfate infusions (given before and after chemotherapy or just before chemotherapy) can prevent or ameliorate chronic, cumulative oxaliplatin-induced sensory neurotoxicity in patients with colon or rectal cancer receiving adjuvant FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin.

Secondary

* To determine whether these 2 infusion schedules can increase the cumulative oxaliplatin doses that can be delivered without dose-limiting chronic neurotoxicity.
* To determine whether these 2 infusion schedules can ameliorate acute neuropathy associated with oxaliplatin.
* To determine whether these 2 infusion schedules cause adverse events.
* To investigate whether these 2 infusions schedules influence patient quality of life.
* To describe baseline and post-treatment neurological quantitative sensory testing abnormalities in the study participants.

Tertiary

* To explore if polymorphisms in the GSTP1, GSTM1, ERCC2, and XRCC1 genes are associated with early onset of oxaliplatin-induced neurotoxicity.

OUTLINE: This is a multicenter study. Patients are stratified according to age (< 65 years vs ≥ 65 years), gender, regimen (FOLFOX4 vs modified FOLFOX6 vs other), and stage of disease (II vs III vs IV). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive calcium gluconate IV and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).
* Arm II: Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).
* Arm III: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).

In all arms, courses repeat every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.

Blood samples are collected before the second course of treatment for translational research.

Patients complete questionnaires on side effects, quality of life, and chemotherapy-induced peripheral neuropathy periodically.

After completion of study treatment, patients are followed up at 3, 6, 12, and 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum
* Has undergone curative resection and is considered to have stage II or III disease or completely resected stage IV disease with no evidence of residual tumor
* Scheduled to receive 6 months of oxaliplatin-based adjuvant chemotherapy with 85 mg/m^2 oxaliplatin every 2 weeks (this includes, for instance, FOLFOX4 or modified FOLFOX6)

  * Patients receiving bevacizumab or cetuximab in combination with FOLFOX as part of a clinical trial or clinical practice are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN
* Serum calcium ≤ 1.2 times ULN
* Serum magnesium ≤ 1.2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to complete questionnaires (alone or with assistance)
* Able to comply with study treatment
* Willing to return to enrolling institution for follow-up
* Willing to provide blood sample for research purposes
* No pre-existing peripheral neuropathy of any grade
* No family history of a genetic/familial neuropathy
* No second or third degree AV heart block or a history of second or third degree heart block

  * Bundle branch blocks are allowed.
* No other medical conditions that, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Central venous access line present, or scheduled to have a central line placed before starting chemotherapy and study treatment
* No prior treatment with neurotoxic chemotherapy (e.g., oxaliplatin, cisplatin, taxanes, or vinca alkaloids)
* No concurrent digitalis medication
* No concurrent treatment with the anticonvulsants carbamazepine (e.g., Tegretol®), phenytoin (e.g., Dilantin®), valproic acid (e.g., Depakene®), gabapentin (Neurontin®), or pregabalin (Lyrica®)
* No concurrent neurotropic agents, including venlafaxine (Effexor), desvenlafaxine (Pristiq®), milnacipran (Savella®), or duloxetine (Cymbalta)
* No concurrent tricyclic antidepressants (such as amitryptilline), or any other agent specifically being given to prevent or treat neuropathy
* No concurrent drugs given as a neuroprotectant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (405):
- United States (404):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kaiser Permanente - Deer Valley, Antioch, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Pismo Beach, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - North Broward Medical Center, Deerfield Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Oncology Center at St. Joseph Hospital, Nashua, New Hampshire
  - Trinitas Comprehensive Cancer Center at Trinitas Hospital, Elizabeth, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Randolph Hospital, Asheboro, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Hematology-Oncology Associates of Fredericksburg, Incorporated, Fredericksburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Hertz DL, Dockter TJ, Satele DV, Loprinzi CL, Le-Rademacher J. Neuropathy severity at the time of oxaliplatin treatment alteration in patients with colon cancer (Alliance A151912). Support Care Cancer. 2021 Dec;29(12):7855-7863. doi: 10.1007/s00520-021-06371-x. Epub 2021 Jun 27. PMID 34176021
- [Derived] Loprinzi CL, Qin R, Dakhil SR, Fehrenbacher L, Flynn KA, Atherton P, Seisler D, Qamar R, Lewis GC, Grothey A. Phase III randomized, placebo-controlled, double-blind study of intravenous calcium and magnesium to prevent oxaliplatin-induced sensory neurotoxicity (N08CB/Alliance). J Clin Oncol. 2014 Apr 1;32(10):997-1005. doi: 10.1200/JCO.2013.52.0536. Epub 2013 Dec 2. PMID 24297951
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium Gluconate + Magnesium Sulfate (Pre and Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).
- Placebo (Pre and Post): Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).
- Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).
Period: Overall Study
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Started (Nine patients were deemed ineligible or withdrew prior to randomization.) | 118 | 119 | 116
Completed | 118 | 119 | 116
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Calcium Gluconate + Magnesium Sulfate (Pre and Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).>>
  >> calcium gluconate: Given IV>>
  >> magnesium sulfate: Given IV>>
  >> oxaliplatin
- Placebo (Pre and Post): Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).>> >> placebo: Given IV>>
  >> oxaliplatin
- Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).>> >> calcium gluconate: Given IV>>
  >> magnesium sulfate: Given IV>>
  >> placebo: Given IV>>
  >>
  >>
  >>> oxaliplatin
- Total: Total of all reporting groups
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post) | Total
Number analyzed (Participants) | 118 | 119 | 116 | 353
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [49 to 65] | 56 [49 to 65] | 57 [50.5 to 64.5] | 56 [50 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 60 | 184
  Male | 56 | 57 | 56 | 169
Region of Enrollment [Count of Participants; unit: Participants]
  Ecuador | 0 | 1 | 0 | 1
  United States | 118 | 118 | 116 | 352

OUTCOME MEASURES:

1. Primary Outcome: Sensory Area Under the Curve(AUC) Score. Oxaliplatin-induced Sensory Neuropathy as Repeatedly Measured by the EORTC QLQ-CIPN20 Sensory Subscale During Chemotherapy
Description: The oxaliplatin-induced sensory neuropathy as repeatedly measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Chemotherapy-induced peripheral neuropathy (EORTC QLQ-CIPN20) sensory subscale during the chemotherapy. This is a multivariate repeated measurement of CIPN with possibly variable cycles for every patient. The CIPN sensory subscale will be calculated by standard scoring algorithm and converted to 0-100 scale, where higher scores represent a higher quality of life. Rather than choosing the CIPN20 sensory subscale at a fixed cycle of chemotherapy, we will adopt a summary measure, area under the curve (AUC) of CIPN20 sensory subscale as the primary endpoint. This AUC will be prorated by the number of chemotherapy cycles patients received.
Time Frame: Up to 18 months
Population: All enrolled patients with Baseline and more than 1 cycle of Sensory data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Calcium Gluconate + Magnesium Sulfate (Pre and Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).>
  >>
  >
  >> calcium gluconate: Given IV>
  >>
  >
  >> magnesium sulfate: Given IV>
  >>
  >
  >> oxaliplatin
- Placebo (Pre and Post): Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).> >>
  >
  >> placebo: Given IV>
  >>
  >
  >> oxaliplatin
- Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).> >>
  >
  >> calcium gluconate: Given IV>
  >>
  >
  >> magnesium sulfate: Given IV>
  >>
  >
  >> placebo: Given IV>
  >>
  >
  >> oxaliplatin
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 110 | 106 | 110
score on a scale | 89.2 (8.5) | 88.3 (9.7) | 87.1 (9.9)
Statistical Analysis 1: Comparison: Calcium Gluconate + Magnesium Sulfate (Pre and Post) vs Placebo (Pre and Post); Two-sample t-tests or Wilcoxon rank-sum tests will be used>> to compare the AUC of CIPN sensory subscale between each of the two schedules of>> Ca/Mg infusions vs placebo arms at the 2.5% significance level. If the CIPN sensory>> subscales are observed to be unbalanced, we will adjust for the baseline CIPN sensory>> subscale scores from the AUC or incorporate them as a covariate in generalized linear>> regression model; Test type: Non-Inferiority or Equivalence — Two-sample t-tests or Wilcoxon rank-sum tests will be used as in>> primary analysis; p = .73, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo (Pre and Post) vs Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Two-sample t-tests or Wilcoxon rank-sum tests will be used as in>> primary analysis; p = .29, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Area Under the Curve (AUC) of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Chemotherapy-induced Peripheral Neuropathy (EORTC QLQ-CIPN20) Autonomic Neuropathy Subscale Scores
Description: The oxaliplatin-induced autonomic neuropathy as repeatedly measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Chemotherapy-induced peripheral neuropathy (EORTC QLQ-CIPN20) autonomic subscale during the chemotherapy. This is a multivariate repeated measurement of CIPN with possibly variable cycles for every patient. The CIPN autonomic subscale will be calculated by standard scoring algorithm and converted to 0-100 scale, where higher scores represent a higher quality of life. Rather than choosing the CIPN20 autonomic subscale at a fixed cycle of chemotherapy, we will adopt a summary measure, area under the curve (AUC) of CIPN20 autonomic subscale as the endpoint. This AUC will be prorated by the number of chemotherapy cycles patients received.
Time Frame: Up to 18 months
Population: All patients with Baseline and more than one cycle of EORTC CIPN-20 Autonomic data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 108 | 102 | 111
score on a scale | 89.8 (12.5) | 86.7 (14.3) | 84.5 (15.1)
Statistical Analysis 1: Comparison: Calcium Gluconate + Magnesium Sulfate (Pre and Post) vs Placebo (Pre and Post); We will not adjust p-values (or significance level) for multiple>> comparisons among the numerous hypothesis testings of secondary endpoints due to the>> exploratory nature of these secondary analyses. The significance results from secondary>> analyses will be interpreted cautiously in a hypothesis-generating fashion; Test type: Non-Inferiority or Equivalence — Two-sample t-tests or Wilcoxon rank-sum tests will be used as in>> primary analysis; p = .054, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo (Pre and Post) vs Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Two-sample t-tests or Wilcoxon rank-sum tests will be used as in>> primary analysis; p = .27, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Area Under the Curve (AUC) of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Chemotherapy-induced Peripheral Neuropathy (EORTC QLQ-CIPN20) Motor Neuropathy Subscale Scores
Description: The oxaliplatin-induced motor neuropathy as repeatedly measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of Chemotherapy-induced peripheral neuropathy (EORTC QLQ-CIPN20) motor neuropathy subscale during the chemotherapy. This is a multivariate repeated measurement of CIPN with possibly variable cycles for every patient. The CIPN motor neuropathy subscale will be calculated by standard scoring algorithm and converted to 0-100 scale, where higher scores represent a higher quality of life. Rather than choosing the CIPN20 motor neuropathy subscale at a fixed cycle of chemotherapy, we will adopt a summary measure, area under the curve (AUC) of CIPN20 motor neuropathy subscale as the endpoint. This AUC will be prorated by the number of chemotherapy cycles patients received.
Time Frame: Up to 18 Months
Population: All patients with at least baseline and more than 1 cycle of Motor Neuropathy data.
Measure: Mean (Standard Deviation); unit: AUC QLQ-CIPN20 Motor Neuropathy Score
Groups:
- Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).>> >> calcium gluconate: Given IV>>
  >> magnesium sulfate: Given IV>>
  >> placebo: Given IV>>
  >> oxaliplatin
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 110 | 106 | 110
AUC QLQ-CIPN20 Motor Neuropathy Score | 94.1 (7.9) | 93.3 (8.0) | 91.6 (10.5)
Statistical Analysis 1: Comparison: Calcium Gluconate + Magnesium Sulfate (Pre and Post) vs Placebo (Pre and Post); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Two-sample t-tests or Wilcoxon rank-sum tests will be used as in>> primary analysis; p = .29, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo (Pre and Post) vs Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post); [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Two-sample t-tests or Wilcoxon rank-sum tests will be used as in>> primary analysis; p = .25, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Patients Experiencing Grade 2+ and Grade 3+ Chronic Cumulative Neurotoxicity.
Description: Grades are determined by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.0) and oxaliplatin-specific neurotoxicity scale, during and after chemotherapy. Higher grades symbolize greater severity of the adverse event.
Time Frame: Up to 18 months
Population: All patients that under went at least one cycle of treatment and were analyzed for chronic cumulative neurotoxicity (NCI CTCAE version 4.0 and oxaliplatin-specific neurotoxicity scale) during and after chemotherapy
Measure: Number; unit: percentage of patients
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 118 | 119 | 116
percentage of patients
  grade 2+ | 42.7 | 44.8 | 46.1
  grade 3+ | 7.7 | 7.8 | 7.8

5. Secondary Outcome: Time to Onset of Grade 2+ and Grade 3+ Chronic Cumulative Neurotoxicity and the Duration of the Chronic Cumulative Neurotoxicity During and After Chemotherapy
Description: Time to onset of grade 2+ and grade 3+ chronic cumulative neurotoxicity, the duration of the chronic cumulative neurotoxicity during and after the adjuvant oxaliplatin-based chemotherapy. Grades are determined by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.0) and oxaliplatin-specific neurotoxicity scale, during and after chemotherapy. Higher grades symbolize greater severity of the adverse event.
Time Frame: Up to 18 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 109 | 108 | 105
Days
  Time to Grade 2 Neuropathy | 171 [154 to 190] | 173 [162 to 181] | 171 [148 to 173]
  Time to Grade 3 Neuropathy | NA [209 to NA] — Not Reached | 208 [200 to NA] — Not Reached | NA [201 to NA] — Not Reached

6. Secondary Outcome: Cumulative Oxaliplatin Doses That Can be Administered Without Dose-limiting Chronic Neurotoxicity
Description: A patient has a dose-limiting chronic neurotoxicity when they discontinue oxaliplatin-based chemotherapy because of neurotoxicity.
Time Frame: Up to 18 months
Population: All patients that discontinued treatment.
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 34 | 32 | 28
Doses | 8.1 (3) | 8.4 (2.5) | 8.0 (2.6)
Statistical Analysis 1: Comparison: Calcium Gluconate + Magnesium Sulfate (Pre and Post) vs Placebo (Pre and Post); Test type: Non-Inferiority or Equivalence — Kruskal Wallis Analysis; p = .89, Kruskal-Wallis
Statistical Analysis 2: Comparison: Placebo (Pre and Post) vs Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post); Test type: Non-Inferiority or Equivalence — Kruskal Wallis Analysis; p = .496, Kruskal-Wallis

7. Secondary Outcome: Percentage of Patients Discontinuing Oxaliplatin-based Chemotherapy Because of Neurotoxicity
Time Frame: Up to 18 months
Population: All patients that received treatment.
Measure: Number; unit: percentage of patients
Groups:
- Calcium Gluconate + Magnesium Sulfate (Pre and Post): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin). >>
  * calcium gluconate: Given IV >>
  * magnesium sulfate: Given IV >>
  * oxaliplatin
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Number analyzed (Participants) | 118 | 119 | 116
percentage of patients | 34.7 | 27.7 | 30.5
Statistical Analysis 1: Comparison: Calcium Gluconate + Magnesium Sulfate (Pre and Post) vs Placebo (Pre and Post); Test type: Non-Inferiority or Equivalence — Chi-Squared Analysis; p = .52, Chi-squared
Statistical Analysis 2: Comparison: Placebo (Pre and Post) vs Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post); Test type: Non-Inferiority or Equivalence — Chi-Squared Analysis; p = .66, Chi-squared

8. Secondary Outcome: Percentage of Patients With Acute Neuropathy Associated With Oxaliplatin
Description: This is the percent of patients who scored >=50 in all sequences of all cycles by arm for side effect Q1: Sensitivity to touching cold. This is a> repeated measurement of CIPN with possibly variable cycles for every patient. The CIPN subscale will be calculated by standard scoring algorithm and converted to 0-100 scale. Where 0 is no sensitivity and 100 is as bad as it can be.
Time Frame: Up to 18 months
Measure: Number; unit: percentage of patients
Groups:
- Arm I: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).>
  >>
  >
  >> calcium gluconate: Given IV>
  >>
  >
  >> magnesium sulfate: Given IV>
  >>
  >
  >> oxaliplatin
- Arm II: Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).> >>
  >
  >> placebo: Given IV>
  >>
  >
  >> oxaliplatin
- Arm III: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).> >>
  >
  >> calcium gluconate: Given IV>
  >>
  >
  >> magnesium sulfate: Given IV>
  >>
  >
  >> placebo: Given IV>
  >>
  >
  >> oxaliplatin
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 110 | 106 | 110
percentage of patients
  Cycle 1 | 10 | 13 | 14
  Cycle 2 | 24 | 27 | 28
  Cycle 3 | 32 | 33 | 32
  Cycle 4 | 34 | 37 | 36
  Cycle 5 | 34 | 33 | 39
  Cycle 6 | 31 | 37 | 33
  Cycle 7 | 35 | 34 | 34
  Cycle 8 | 32 | 34 | 33
  Cycle 9 | 34 | 37 | 32
  Cycle 10 | 29 | 39 | 30
  Cycle 11 | 28 | 39 | 33
  Cycle 12 | 27 | 45 | 32

9. Secondary Outcome: Incidence of Calcium Gluconate and Magnesium Sulfate-induced Adverse Events as Measured by CTCAE Version 4.0
Time Frame: Up to 18 months
Measure: Number; unit: Number of reported Adverse Events
Groups:
- Arm I: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy comprising leucovorin calcium, fluorouracil, and oxaliplatin).>>
  >> calcium gluconate: Given IV>>
  >> magnesium sulfate: Given IV>>
  >> oxaliplatin
- Arm II: Patients receive placebo IV over 30 minutes immediately before and after oxaliplatin administration (part of FOLFOX chemotherapy).>> >> placebo: Given IV>>
  >> oxaliplatin
- Arm III: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and placebo IV over 30 minutes immediately after oxaliplatin administration (part of FOLFOX chemotherapy).>> >> calcium gluconate: Given IV>>
  >> magnesium sulfate: Given IV>>
  >> placebo: Given IV>>
  >> oxaliplatin
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 118 | 119 | 116
Number of reported Adverse Events | 290 | 259 | 296

10. Secondary Outcome: Area Under the Curve (AUC) of Patient-reported Quality of Life (QOL) as Measured by the Supplemental QOL Questionnaire
Description: This is a multivariate repeated measurement of CIPN with possibly variable cycles for every patient. The supplemental quality of life (QOL) subscale will be calculated by standard scoring algorithm and converted to 0-100 scale, where higher scores represent a higher quality of life. Rather than choosing the subscale at a fixed cycle of chemotherapy, we will adopt a summary measure, area under the curve (AUC) . This AUC will be prorated by the number of chemotherapy cycles patients received.
Time Frame: Up to 18 months
Population: All patients that had at least one cycle of treatment and submitted a patient-reported quality of life (QOL) as measured by the supplemental QOL questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I | Arm II | Arm III
Number analyzed (Participants) | 111 | 112 | 108
score on a scale
  Diarrhea | 86.7 (15.5) | 86.2 (15.7) | 84.5 (16)
  Constipation | 90.1 (13.0) | 88.8 (13.4) | 88.0 (18.8)
  Stomach Cramping | 92.8 (11.4) | 90.6 (12.6) | 89.4 (15.6)
  Bowel Problems | 89.1 (13.4) | 88.5 (14.4) | 84.6 (19.0)
  Swallowing | 91.2 (10.0) | 87.6 (13.8) | 86.7 (14.1)
  Numbness in finger and toes | 83.4 (14.8) | 81.8 (15.7) | 80.0 (17.3)
  Tingling in finger and toes | 78.9 (16.5) | 76.5 (17.3) | 76.3 (17.6)

ADVERSE EVENTS:
Time Frame: 3 years
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for adverse event monitoring and reporting. The CTCAE version 4.0 can be accessed from the CTEP home page (http://ctep.cancer.gov).
Groups:
- Calcium Gluconate + Magnesium Sulfate (Pre and Post); Placebo (Pre and Post); Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post): oxaliplatin
Arm/Group | Calcium Gluconate + Magnesium Sulfate (Pre and Post) | Placebo (Pre and Post) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post)
Serious Adverse Events (participants affected / at risk) | 13/117 | 9/119 | 8/116
Other Adverse Events (participants affected / at risk) | 107/117 | 108/119 | 105/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Gluconate + Magnesium Sulfate (Pre and Post) (N=117) | Placebo (Pre and Post) (N=119) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post) (N=116)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (13) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0) | 3 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (4) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Gluconate + Magnesium Sulfate (Pre and Post) (N=117) | Placebo (Pre and Post) (N=119) | Calcium Gluconate + Magnesium Sulfate (Pre), Placebo (Post) (N=116)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 2 (7) | 4 (6)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 4 (4) | 4 (4)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 3 (14) | 2 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 4 (8) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 80 (315) | 73 (325) | 77 (363)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 5 (5) | 4 (5)
Nausea (Gastrointestinal disorders) | 86 (351) | 78 (346) | 78 (377)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 42 (70) | 30 (55) | 33 (84)
Fatigue (General disorders) | 9 (22) | 13 (32) | 13 (30)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 2 (9) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (9) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 2 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 28 (54) | 28 (51) | 32 (67)
Platelet count decreased (Investigations) | 8 (18) | 8 (15) | 8 (16)
Weight gain (Investigations) | 1 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 13 (20) | 10 (17) | 14 (21)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (5) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 2 (3) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 14 (33) | 12 (23) | 10 (18)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (4)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (8) | 3 (4) | 2 (9)
Hypotension (Vascular disorders) | 2 (2) | 3 (3) | 2 (2)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (14) | 3 (4) | 5 (10)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes